CLINICAL TRIAL: NCT04640350
Title: Risk Prediction of Bleeding in Liver Cirrhosis by Combi-elastography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Chinese PLA General Hospital
Other Study IDs: S2020-387-02
Record Dates: First submitted 2020-11-10; First posted 2020-11-23 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Liver Cirrhosis; Gastroesophageal Varices; Variceal Hemorrhage
Keywords: Elasticity Imaging Techniques; Ultrasound
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through the parameters of liver stiffness and spleen stiffness obtained by combi-elastography technique, summarize and analyze the warning index of esophagogastric variceal bleeding in patients with cirrhosis, so as to provide a new and valuable technique for clinical diagnosis.

DETAILED DESCRIPTION:
Firstly,the combi-elastography technique developed by HITACHI uses the method of multi-index and multi-parameter to evaluate the liver stiffness and spleen stiffness comprehensively.

And then,this prospective study is designed to follow up patients with cirrhosis for a period of 12 months, summarize and analyze the warning index of bleeding in patients with cirrhosis,so as to provide a new and valuable technique for clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old, no gender limit;
* The clinical diagnosis is in line with patients with liver cirrhosis caused by chronic hepatitis B, and the gastroscopy is in line with the indications of portal hypertension;
* Gastroscopy needs to provide the degree of gastroesophageal varices;
* Sign the informed consent form.

Exclusion Criteria:

* Patients with cirrhosis and portal hypertension because of other causes or combined with other causes(such as viral hepatitis other than hepatitis B,Autoimmune liver disease, alcoholic liver disease, metabolism-related fatty liver disease, etc.)
* Patients with a history of spleen-related operations, such as splenectomy, splenic embolism;
* Patients undergoing portosystemic shunt or TIPS;
* Isolated esophageal venous tumor and its bleeding patients;
* History of upper gastrointestinal tumor or bleeding from gastric ulcer , etc;
* Those with serious diseases of other systems that cannot cooperate with elastography examination, such as heart failure, renal failure, mental illness, etc;
* Ascites before liver and spleen result unable to complete elasticity examination;
* Pregnant patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis and the gastroscopy is in line with the indications of portal hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
F index | baseline
  F index is linked to the degree of liver fibrosis,and it can be available by ultrasound elastography checking.
A index | baseline
  A index is linked to the degree of hepatitis ,and it can be available by ultrasound elastography checking.
Spleen stiffness | baseline
  Spleen stiffness can be available by ultrasound elastography checking.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China